CLINICAL TRIAL: NCT03607097
Title: Integral Management of Healthcare Problems Related With Drugs in Polimedicated Patients: Drug Code
Brief Title: Integral Management of Healthcare Problems Related With Drugs in Polimedicated Patients: Medication Code
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIBSP-COD-2018-25
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Drug Related Problems; Pharmaceutical Care
Keywords: secondary prevention; pharmaceutical care; drug related problems; emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secondary prevention of DRPs (medication code) (intervention) (Experimental): The intervention consists of :1)Patient-centred prescription Espaulella-Panicot J model (review model that includes different strategies in a single intervention. It is performed by a multidisciplinary team, and allows them to adapt the pharmacological plan of patients with clinical complexity). 2)strategies to improve medication adherence
  Interventions: Procedure: Secondary prevention program for drug related problems
- Usual care (control group) (No Intervention): The patient is reviewed according to the standard procedure, consisting only on the review of the medical prescription in the emergency department by the pharmacist assisting the unit

INTERVENTIONS:
Procedure: Secondary prevention program for drug related problems — The interventions consists of three stages: 1) actions aimed at improving the chronic prescription of the patient, 2) actions aimed at improving the therapeutic adherence and 3) actions aimed at improving the assistance healthcare levels coordination
  Other Names: Medication Code
  Arms: Secondary prevention of DRPs (medication code) (intervention)

SUMMARY:
Background:

Although Drug- related Problems (DRPs) in polimedicated patients are a major public health problem in western countries and many of them have been considered avoidable, secondary and primary prevention policies have not been systematized, beyond pharmaceutical care programs in certain settings and on specific patients.

Objectives:

The main objective of this study is to evaluate the impact of implementing the Medication Code (CM) on patients who consult the emergency department for a DRP (secondary prevention of DRP). It is also intended to draw conclusions, based on the knowledge obtained in terms of DRP that will allow the establishment of future actions to reduce its prevalence (primary prevention actions).

Method:

A single-centre clinical trial is proposed in which adult patients will be selected to consult the Hospital Emergency Department (ED) of the Hospital de la Santa Creu i Sant Pau (HSCSP) for a primary or secondary diagnosis of DRP and will be randomised with a 1:1 distribution to be included in the medication code (intervention group) or to receive usual care (control group). The intervention will be evaluated in terms of health outcomes (ED consultations and hospital readmission).

DETAILED DESCRIPTION:
A single-centre clinical trial is proposed in which adult patients will be selected to consult the Hospital Emergency Department (ED) of the Hospital de la Santa Creu i Sant Pau (HSCSP) for a primary or secondary diagnosis of DRP and will be randomised with a 1:1 distribution to be included in the medication code (intervention group) or to receive usual care (control group). The intervention will be evaluated in terms of health outcomes (ED consultations and hospital readmission).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Drug Related Problems (DRP) related to drugs from Anatomical Therapeutic Chemical (ATC) groups A, B and C

Exclusion Criteria:

* DRP due to autolytic attempt or final phase of life.
* Denied informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
30 day readmission | 30 days
  Readmissions during the 30 days after the intervention in any hospital centre from the "Àrea Integral de Salut Barcelona Dreta" after consulting the Hospital de la Santa Creu i Sant Pau (HSCSP) emergency department.

SECONDARY OUTCOMES:
30 day consultation | 30 days
  Consultation 30 days after the intervention for any cause to the HSCSP
30 day mortality | 30 days
  Any cause mortality 30 days after the intervention
Time on Emergency Department | 72 hours
  Time from patient admission to discharge from the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Juanes, PhD, Principal Investigator — Hospital Sante Creu i Sant Pau, Barcelona (Spain)
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Background] Nivya K, Sri Sai Kiran V, Ragoo N, Jayaprakash B, Sonal Sekhar M. Systemic review on drug related hospital admissions - A pubmed based search. Saudi Pharm J. 2015 Jan;23(1):1-8. doi: 10.1016/j.jsps.2013.05.006. Epub 2013 May 30. PMID 25685036
- [Background] Baena MI, Fajardo PC, Pintor-Marmol A, Faus MJ, Marin R, Zarzuelo A, Martinez-Olmos J, Martinez-Martinez F. Negative clinical outcomes of medication resulting in emergency department visits. Eur J Clin Pharmacol. 2014 Jan;70(1):79-87. doi: 10.1007/s00228-013-1562-0. Epub 2013 Oct 3. PMID 24091839
- [Background] Castro I, Guardiola JM, Tuneu L, Sala ML, Faus MJ, Mangues MA. Drug-related visits to the emergency department in a Spanish university hospital. Int J Clin Pharm. 2013 Oct;35(5):727-35. doi: 10.1007/s11096-013-9795-7. Epub 2013 May 22. PMID 23695594
- [Background] Patel P, Zed PJ. Drug-related visits to the emergency department: how big is the problem? Pharmacotherapy. 2002 Jul;22(7):915-23. doi: 10.1592/phco.22.11.915.33630. PMID 12126224
- [Background] Queneau P, Bannwarth B, Carpentier F, Guliana JM, Bouget J, Trombert B, Leverve X, Lapostolle F, Borron SW, Adnet F; Association Pedagogique Nationale pour l'Enseignement de la Therapeutique (APNET). Emergency department visits caused by adverse drug events: results of a French survey. Drug Saf. 2007;30(1):81-8. doi: 10.2165/00002018-200730010-00008. PMID 17194173
- [Background] Wei L, Yang X, Li J, Liu L, Luo H, Zheng Z, Wei Y. Effect of pharmaceutical care on medication adherence and hospital admission in patients with chronic obstructive pulmonary disease (COPD): a randomized controlled study. J Thorac Dis. 2014 Jun;6(6):656-62. doi: 10.3978/j.issn.2072-1439.2014.06.20. PMID 24976987
- [Background] Obreli-Neto PR, Marusic S, Guidoni CM, Baldoni Ade O, Renovato RD, Pilger D, Cuman RK, Pereira LR. Economic evaluation of a pharmaceutical care program for elderly diabetic and hypertensive patients in primary health care: a 36-month randomized controlled clinical trial. J Manag Care Spec Pharm. 2015 Jan;21(1):66-75. doi: 10.18553/jmcp.2015.21.1.66. PMID 25562774
- [Background] Koshman SL, Charrois TL, Simpson SH, McAlister FA, Tsuyuki RT. Pharmacist care of patients with heart failure: a systematic review of randomized trials. Arch Intern Med. 2008 Apr 14;168(7):687-94. doi: 10.1001/archinte.168.7.687. PMID 18413550
- [Background] Ravn-Nielsen LV, Duckert ML, Lund ML, Henriksen JP, Nielsen ML, Eriksen CS, Buck TC, Pottegard A, Hansen MR, Hallas J. Effect of an In-Hospital Multifaceted Clinical Pharmacist Intervention on the Risk of Readmission: A Randomized Clinical Trial. JAMA Intern Med. 2018 Mar 1;178(3):375-382. doi: 10.1001/jamainternmed.2017.8274. PMID 29379953
- [Derived] Juanes A, Ruiz J, Puig M, Blazquez M, Gilabert A, Lopez L, Baena MI, Guiu JM, Antonia Mangues M. The Effect of the Drug-Related Problems Prevention Bundle on Early Readmissions in Patients From the Emergency Department: A Randomized Clinical Trial. Ann Pharmacother. 2023 Sep;57(9):1025-1035. doi: 10.1177/10600280221143237. Epub 2022 Dec 20. PMID 36539949